CLINICAL TRIAL: NCT01297127
Title: Prospective Multicentre Noninterventional Observational Study on Predictors of Treatment Response in a Cohort of Treatment naïve HIV-infected Patients Treated With Saquinavir (PROSPECTOR)
Brief Title: Observational Study on Predictors of Response to Invirase (Saquinavir) Treatment in Treatment-naïve Patients With HIV Infection
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25398
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective observational study will evaluate predictors of response to Invirase (saquinavir) treatment in treatment-naïve patients with HIV infection. Data will be collected during 48 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* HIV infection
* Treatment-naïve
* Initiation of treatment with Invirase

Exclusion Criteria:

* Contraindications according to Invirase Summary of Product Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment-naïve HIV-infected patients initiated on treatment with Invirase
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2010-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Predictive value of baseline CD4 count and HIV RNA on virological and immunological response at 12, 24 and 48 weeks of treatment | 48 weeks

SECONDARY OUTCOMES:
Host- and virus-related factors influencing virological and immunological response at 12, 24 and 48 weeks of treatment | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Poland (8):
  - Bialystok
  - Bydgoszcz
  - Chorzów
  - Krakow
  - Lodz
  - Warsaw
  - Wroclaw
  - Zielona Góra